CLINICAL TRIAL: NCT04033146
Title: Optimizing Ankle Exoskeleton Assistance for Walking Across the Life Span
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H18208; F32AG063460 (NIH)
Record Dates: First submitted 2019-07-23; First posted 2019-07-25 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Aging
Keywords: Walking; Aging; Exoskeleton Device

STUDY DESIGN:
Intervention Model Description: All participants will perform the same trials/sessions to complete the entire protocol. After each participant has performed all trials for this study, the investigators will analyze the data of this repeated-measures design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Young Adult Exoskeleton Users (Experimental): Study participants who are 18-45 year old.
  Interventions: Device: Ankle Exoskeleton Assistance
- Older Adult Exoskeleton Users (Experimental): Study participants who are greater than 65 years of age.
  Interventions: Device: Ankle Exoskeleton Assistance

INTERVENTIONS:
Device: Ankle Exoskeleton Assistance — The investigators will use ankle-exoskeletons to modulate the amount of mechanical power generated by the user's ankle joint. That is, participants will walk in a robotic device that either (a) adds a spring or (b) a motor in parallel with their calf muscles to help them generate a stronger propulsive push-off that could reduce the effort of walking.

SUMMARY:
The investigators seek to determine whether ankle exoskeletons can reduce metabolic energy expenditure during walking for users across the age-spectrum.

DETAILED DESCRIPTION:
Older adults walk with greater metabolic rates than young adults. Growing evidence suggests that the greater older adult metabolic rates are related to the structural properties of their lower leg tissues. The tendons of the leg of older adults are more compliant than that of young adults. Accordingly, older adult leg tendons stretch more under a given load, such as during walking, causing their muscles to operate at shorter, less optimal lengths, and higher activity levels than the muscles of young adults - a less economical way to produces force.

Thus, the investigators seek to examine whether wearing wearable robotic boots (i.e., ankle exoskeletons) could enable muscles to produce force more economically. By adding an exoskeleton in-parallel to the ankle, the investigators hypothesize that older adults will walk with lower whole-body metabolic rate than without the exoskeleton assistance.

In this study, the investigators will have both young and older adult participants walk on a treadmill with a commercially available ankle exoskeleton set in multiple assistance modes. During these trials, the investigators will measure the metabolic cost of walking in young and older adults and also take many physiological and biomechanical measurements to help assess how exoskeletons work to reduce walking effort.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to walk for 60 minutes in a 90-minute time frame.
* Subjects are apparently free of cardiovascular, metabolic, and renal disease, which includes no signs or symptoms suggestive of cardiovascular, metabolic or renal disease.
* Subjects have no current musculoskeletal injury.
* Subjects need to be either 18-45 or 65+ years old.

These criteria meet the American College of Sports Medicine's 2015 guidelines for participant health screening prior to joining a moderate or moderate-to-vigorous exercise protocol. (Riebe et al., 2015).

Exclusion Criteria:

* Have dementia or an inability to give informed consent
* Have a musculoskeletal injury or feel pain while walking
* Have a history of dizziness and/or balance problems
* Have cardiovascular, heart, metabolic, or renal disease, or respiratory problems
* Smoke cigarettes
* Asthma
* Feel pain or discomfort in the chest, neck, jaw, arms during rest or exercise
* Have orthopnea or paroxysmal nocturnal dyspnea
* Have ankle edema
* Have palpitations or tachycardia
* Have a heart murmur
* Have had a heart attack
* Have diabetes
* Have a pace maker
* Have unusual shortness of breath with usual activities
* Are <18 or 46-64 years of age
* Do not speak or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory S Sawicki, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Physiology of Wearable Robotics Laboratory (Georgia Tech), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asbeck AT, De Rossi SM, Holt KG, and Walsh CJ. A biologically inspired soft exosuit for walking assistance. The international journal of robotics research 34: 744-762, 2015.
- [Background] Biewener AA, Farley CT, Roberts TJ, Temaner M. Muscle mechanical advantage of human walking and running: implications for energy cost. J Appl Physiol (1985). 2004 Dec;97(6):2266-74. doi: 10.1152/japplphysiol.00003.2004. Epub 2004 Jul 16. PMID 15258124
- [Background] Browne MG, Franz JR. The independent effects of speed and propulsive force on joint power generation in walking. J Biomech. 2017 Apr 11;55:48-55. doi: 10.1016/j.jbiomech.2017.02.011. Epub 2017 Feb 21. PMID 28262285
- [Background] Cavagna GA, Kaneko M. Mechanical work and efficiency in level walking and running. J Physiol. 1977 Jun;268(2):467--81. doi: 10.1113/jphysiol.1977.sp011866. PMID 874922
- [Background] CAVAGNA GA, SAIBENE FP, MARGARIA R. MECHANICAL WORK IN RUNNING. J Appl Physiol. 1964 Mar;19:249-56. doi: 10.1152/jappl.1964.19.2.249. No abstract available. PMID 14155290
- [Background] Collins SH, Wiggin MB, Sawicki GS. Reducing the energy cost of human walking using an unpowered exoskeleton. Nature. 2015 Jun 11;522(7555):212-5. doi: 10.1038/nature14288. Epub 2015 Apr 1. PMID 25830889
- [Background] Csapo R, Malis V, Hodgson J, Sinha S. Age-related greater Achilles tendon compliance is not associated with larger plantar flexor muscle fascicle strains in senior women. J Appl Physiol (1985). 2014 Apr 15;116(8):961-9. doi: 10.1152/japplphysiol.01337.2013. Epub 2014 Feb 6. PMID 24505104
- [Background] DeVita P, Helseth J, Hortobagyi T. Muscles do more positive than negative work in human locomotion. J Exp Biol. 2007 Oct;210(Pt 19):3361-73. doi: 10.1242/jeb.003970. PMID 17872990
- [Background] DeVita P, Hortobagyi T. Age causes a redistribution of joint torques and powers during gait. J Appl Physiol (1985). 2000 May;88(5):1804-11. doi: 10.1152/jappl.2000.88.5.1804. PMID 10797145
- [Background] Elliott G, Sawicki GS, Marecki A, Herr H. The biomechanics and energetics of human running using an elastic knee exoskeleton. IEEE Int Conf Rehabil Robot. 2013 Jun;2013:6650418. doi: 10.1109/ICORR.2013.6650418. PMID 24187237
- [Background] Farris DJ, Sawicki GS. The mechanics and energetics of human walking and running: a joint level perspective. J R Soc Interface. 2012 Jan 7;9(66):110-8. doi: 10.1098/rsif.2011.0182. Epub 2011 May 25. PMID 21613286
- [Background] Ferris DP, Sawicki GS, Domingo A. Powered lower limb orthoses for gait rehabilitation. Top Spinal Cord Inj Rehabil. 2005;11(2):34-49. doi: 10.1310/6gl4-um7x-519h-9jyd. PMID 16568153
- [Background] Franz JR, Slane LC, Rasske K, Thelen DG. Non-uniform in vivo deformations of the human Achilles tendon during walking. Gait Posture. 2015 Jan;41(1):192-7. doi: 10.1016/j.gaitpost.2014.10.001. Epub 2014 Oct 12. PMID 25457482
- [Background] Gottschall JS, Kram R. Energy cost and muscular activity required for propulsion during walking. J Appl Physiol (1985). 2003 May;94(5):1766-72. doi: 10.1152/japplphysiol.00670.2002. Epub 2002 Dec 27. PMID 12506042
- [Background] Griffin TM, Tolani NA, Kram R. Walking in simulated reduced gravity: mechanical energy fluctuations and exchange. J Appl Physiol (1985). 1999 Jan;86(1):383-90. doi: 10.1152/jappl.1999.86.1.383. PMID 9887153
- [Background] Holt NC, Roberts TJ, Askew GN. The energetic benefits of tendon springs in running: is the reduction of muscle work important? J Exp Biol. 2014 Dec 15;217(Pt 24):4365-71. doi: 10.1242/jeb.112813. Epub 2014 Nov 13. PMID 25394624
- [Background] Huang HJ, Kram R, Ahmed AA. Reduction of metabolic cost during motor learning of arm reaching dynamics. J Neurosci. 2012 Feb 8;32(6):2182-90. doi: 10.1523/JNEUROSCI.4003-11.2012. PMID 22323730
- [Background] Malcolm P, Derave W, Galle S, De Clercq D. A simple exoskeleton that assists plantarflexion can reduce the metabolic cost of human walking. PLoS One. 2013;8(2):e56137. doi: 10.1371/journal.pone.0056137. Epub 2013 Feb 13. PMID 23418524
- [Background] Martin PE, Rothstein DE, Larish DD. Effects of age and physical activity status on the speed-aerobic demand relationship of walking. J Appl Physiol (1985). 1992 Jul;73(1):200-6. doi: 10.1152/jappl.1992.73.1.200. PMID 1506370
- [Background] Mian OS, Thom JM, Ardigo LP, Minetti AE, Narici MV. Gastrocnemius muscle-tendon behaviour during walking in young and older adults. Acta Physiol (Oxf). 2007 Jan;189(1):57-65. doi: 10.1111/j.1748-1716.2006.01634.x. PMID 17280557
- [Background] Mooney LM, Rouse EJ, Herr HM. Autonomous exoskeleton reduces metabolic cost of human walking during load carriage. J Neuroeng Rehabil. 2014 May 9;11:80. doi: 10.1186/1743-0003-11-80. PMID 24885527
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Nuckols Rich DT, Sawicki Greg. Ultrasound measurements link soleus muscle dynamics and metabolic cost during human walking with elastic ankle exoskeletons. In Prep.
- [Background] Onambele GL, Narici MV, Maganaris CN. Calf muscle-tendon properties and postural balance in old age. J Appl Physiol (1985). 2006 Jun;100(6):2048-56. doi: 10.1152/japplphysiol.01442.2005. Epub 2006 Feb 2. PMID 16455811
- [Background] Ortega JD, Beck ON, Roby JM, Turney AL, Kram R. Running for exercise mitigates age-related deterioration of walking economy. PLoS One. 2014 Nov 20;9(11):e113471. doi: 10.1371/journal.pone.0113471. eCollection 2014. PMID 25411850
- [Background] Ortega JD, Farley CT. Individual limb work does not explain the greater metabolic cost of walking in elderly adults. J Appl Physiol (1985). 2007 Jun;102(6):2266-73. doi: 10.1152/japplphysiol.00583.2006. Epub 2007 Mar 15. PMID 17363623
- [Background] Ortega JO, Lindstedt SL, Nelson FE, Jubrias SA, Kushmerick MJ, Conley KE. Muscle force, work and cost: a novel technique to revisit the Fenn effect. J Exp Biol. 2015 Jul;218(Pt 13):2075-82. doi: 10.1242/jeb.114512. Epub 2015 May 11. PMID 25964423
- [Background] Panizzolo FA, Green DJ, Lloyd DG, Maiorana AJ, Rubenson J. Soleus fascicle length changes are conserved between young and old adults at their preferred walking speed. Gait Posture. 2013 Sep;38(4):764-9. doi: 10.1016/j.gaitpost.2013.03.021. Epub 2013 May 1. PMID 23642629
- [Background] Rall JA. Sense and nonsense about the Fenn effect. Am J Physiol. 1982 Jan;242(1):H1-6. doi: 10.1152/ajpheart.1982.242.1.H1. PMID 7058903
- [Background] Rasske K, Thelen DG, Franz JR. Variation in the human Achilles tendon moment arm during walking. Comput Methods Biomech Biomed Engin. 2017 Feb;20(2):201-205. doi: 10.1080/10255842.2016.1213818. Epub 2016 Jul 27. PMID 27460018
- [Background] Rubenson J, Pires NJ, Loi HO, Pinniger GJ, Shannon DG. On the ascent: the soleus operating length is conserved to the ascending limb of the force-length curve across gait mechanics in humans. J Exp Biol. 2012 Oct 15;215(Pt 20):3539-51. doi: 10.1242/jeb.070466. Epub 2012 Jul 5. PMID 22771749
- [Background] Sawicki GS, Ferris DP. Mechanics and energetics of level walking with powered ankle exoskeletons. J Exp Biol. 2008 May;211(Pt 9):1402-13. doi: 10.1242/jeb.009241. PMID 18424674
- [Background] Stanaway FF, Gnjidic D, Blyth FM, Le Couteur DG, Naganathan V, Waite L, Seibel MJ, Handelsman DJ, Sambrook PN, Cumming RG. How fast does the Grim Reaper walk? Receiver operating characteristics curve analysis in healthy men aged 70 and over. BMJ. 2011 Dec 15;343:d7679. doi: 10.1136/bmj.d7679. PMID 22174324
- [Background] Stenroth L, Peltonen J, Cronin NJ, Sipila S, Finni T. Age-related differences in Achilles tendon properties and triceps surae muscle architecture in vivo. J Appl Physiol (1985). 2012 Nov;113(10):1537-44. doi: 10.1152/japplphysiol.00782.2012. Epub 2012 Oct 4. PMID 23042907
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Background] Takahashi KZ, Gross MT, van Werkhoven H, Piazza SJ, Sawicki GS. Adding Stiffness to the Foot Modulates Soleus Force-Velocity Behaviour during Human Walking. Sci Rep. 2016 Jul 15;6:29870. doi: 10.1038/srep29870. PMID 27417976
- [Background] Takahashi KZ, Lewek MD, Sawicki GS. A neuromechanics-based powered ankle exoskeleton to assist walking post-stroke: a feasibility study. J Neuroeng Rehabil. 2015 Feb 25;12:23. doi: 10.1186/s12984-015-0015-7. PMID 25889283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled and participated in the study from 2/4/2020 to 5/23/2023.
Groups:
- Older Adult Exoskeleton Users: Study participants who are >65 years old
Period: Overall Study
Arm/Group | Young Adult Exoskeleton Users | Older Adult Exoskeleton Users
Started | 10 | 6
Completed | 10 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Adult Exoskeleton Users | Older Adult Exoskeleton Users | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 6 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 7 | 1 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Net Metabolic Rate (Watts/kg)
Description: The rate of metabolic energy that participants expend during a short walking bout in each of the experimental conditions.
Time Frame: 3rd session, up to 2 weeks
Measure: Mean (Standard Deviation); unit: watts/kg
Arm/Group | Young Adult Exoskeleton Users | Older Adult Exoskeleton Users
Number analyzed (Participants) | 10 | 6
watts/kg
  No Exoskeleton | 3.30 (0.66) | 3.47 (0.31)
  No Torque | 3.86 (0.62) | 4.18 (0.62)
  Spring-like Torque | 3.72 (0.78) | 4.34 (0.57)
  Motor-like Low Torque | 3.51 (0.83) | 3.68 (0.65)
  Motor-like Medium Torque | 3.13 (0.70) | 3.46 (0.56)
  Motor-like High Torque | 3.24 (0.65) | 3.20 (0.52)
Statistical Analysis 1: Comparison: Young Adult Exoskeleton Users vs Older Adult Exoskeleton Users; H1. Bilateral ankle exoskeletons that provide 'motor-like' assistance will result in lower net metabolic power than those providing 'spring-like' assistance for young adults. H2. Bilateral ankle exoskeletons that provide 'motor-like' assistance will result in lower net metabolic power than those providing 'spring-like' assistance for older adults; Test type: Other; p < 0.001, ANOVA — Threshold was 0.05

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Young Adult Exoskeleton Users | Older Adult Exoskeleton Users
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 0/10 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04033146/Prot_001.pdf
  • Statistical Analysis Plan (2024-04-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT04033146/SAP_002.pdf
  • Informed Consent Form (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/46/NCT04033146/ICF_000.pdf